CLINICAL TRIAL: NCT04372446
Title: Understanding the Spectrum of ENPP1 Deficiency and Acute ABCC6 Deficiency Through the Eyes of Patients and Parents; Burden of Illness Perspectives From Patients and Parents Who Speak English, French or German
Brief Title: Understanding the Spectrum of ENPP1 Deficiency and Acute ABCC6 Deficiency
Status: Completed | Type: Observational
Sponsor: Inozyme Pharma (Industry)
Collaborators: GACI Global (Unknown); Engage Health Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: INZ701-004
Record Dates: First submitted 2020-04-13; First posted 2020-05-04 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Generalized Arterial Calcification in Infancy; Autosomal Recessive Hypophosphatemic Rickets Type 2
Keywords: ENPP1 deficiency and ABCC6 deficiency
MeSH Terms: conditions — Arterial calcification of infancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To date, the investigators lack characterization of, the burden of, and the systemic progression of disease in ENPP1 deficiency and ABCC6 deficiency from a patient and/or parent perspective. This study aims to document this characterization, progression as well as the burden of disease. Link to the study registration-

https://www.engagehealth.com/survey/TakeSurvey.aspx?SurveyID=8252n62

DETAILED DESCRIPTION:
This will be a comprehensive, cross-sectional study conducted in approximately 60 individuals (or representative parents of patients) affected by ENPP1 deficiency and the acute form of ABCC6 deficiency. All study participants will complete the RSVP, PRO tools and upload a proof of disease form, followed by an interview conducted by a trained interviewer. It is estimated that each respondent will need up to 60 minutes for the entire process; 20 minutes to complete the RSVP, PRO tools and to upload proof of diagnosis of ENPP1 deficiency or the acute form of ABBC6 deficiency, and approximately 40 minutes to complete the interview and address any follow-up questions if needed.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be a person with ENPP1 deficiency or the acute infantile form of ABCC6 deficiency who is 18 years or older
2. The parent/caregiver of a patient who has been diagnosed with ENPP1 deficiency or the acute infantile form of ABCC6 deficiency. Please note, parents/caregivers of patients with ENPP1 deficiency who have passed away may participate
3. Confirmed diagnosis of ENPP1 deficiency or ABCC6 deficiency with written proof of disease provided
4. Ability to participate in the RSVP and interview in German, French or English, irrespective of country of residence.
5. Able to grant informed consent
6. Willing to participate in a 40-to-60-minute telephone interview, including follow up questions (if necessary)

Exclusion Criteria:

* Inability to meet any of the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 60 participants across four groups; person or parent/legal guardian affected by ENPP1 (GACI or ARHR2) or the acute form of ABCC6 def. described below;
  * Acute infantile ENPP1 def. (due to the high infant mortality, this group likely to include parents of affected children, both living and deceased)
  * Acute infantile ABCC6 def. (due to the high infant mortality, this group likely to include parents of affected children, both living and deceased)
  * Progressive pediatric ENPP1 def. who are still growing (note; due to the age of those who are still growing, this group is likely to include parents of affected children)
  * Adult ENPP1 def. who are no longer growing (note: due to the age of those who are no longer growing, this group is likely to include both patients > age 18 years and parents of affected children who are < age 18 years or who are unable to answer for themselves)
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
To improve the understanding of the characterization and burden of disease in ENPP1 deficient, and acute ABCC6 deficient, patients who are still growing and those who are done growing | Data will be collected during a 45 minute interview. This will be a patient or parent report of events that occurred from birth to the patient's current age which will differ for all respondents.
  The burden of disease through the eyes/voice of the patient and or caregiver will be collected and analyze for improved understanding
To collect information regarding disease burden, in the patient's / families own terms | Data will be collected during a 45 minute interview. This will be a patient or parent report of events that occurred from birth to the patient's current age which will differ for all respondents.
  Data will be collected in terms used by the patient and or caregiver
To build a foundation of evidence to contribute to the dossier, used for many purposes, including reimbursement and regulatory bodies. | Data will be collected during a 45 minute interview. This will be a patient or parent report of events that occurred from birth to the patient's current age which will differ for all respondents.
  Data will be collected and analyzed to be able to draw meaningful conclusions regarding burden of disease in the voice of patients and caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Huertas, MD, Principal Investigator — Inozyme Pharma
Locations (1):
- Engage Health, Eagan, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Registration link to participate in the survey — http://www.engagehealth.com/survey/TakeSurvey.aspx?SurveyID=8252n62

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT04372446/Prot_SAP_000.pdf